CLINICAL TRIAL: NCT00596661
Title: A Prospective, Multi-Center, Non-Randomized, Single-Arm Trial to Evaluate the Safety and Feasibility of the TriMaxx Coronary Stent in de Novo Coronary Artery Lesions.
Brief Title: The TRIMAXX Coronary Stent Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Manager Medical Information, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVD 640-0051-01
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TRIMAXX (Experimental): TRIMAXX Coronary Stent
  Interventions: Device: TriMaxx Coronary Stent placement

INTERVENTIONS:
Device: TriMaxx Coronary Stent placement — Angioplasty with coronary artery stent placement
  Other Names: TriMaxx™ Coronary Stent

SUMMARY:
The primary objective of the trial is to demonstrate the safety and feasibility of treating coronary artery lesions which have not been previously treated with the TRIMAXX Coronary stent system as compared to the reported results for commercially available non-drug eluting coronary stent systems which are indicated for the same treatments.

DETAILED DESCRIPTION:
The TriMaxx study is a prospective, multicenter, non-randomized, single-arm trial intended to demonstrate the safety and feasibility of the TriMaxx Cornary Stent System. The study will enroll 100 subjects with de novo native coronary artery lesions who meet the eligibility criteria and agree to participate in the study. Subjects will be enrolled in a sequential manner. The safety and feasibility of the TRIMAXX stent will be evaluated by comparing the MACE rate that is observed 30 days post-procedure to the MACE rate for commercially available non-drug eluting stents. Secoandry evaluations will include analysis of clinical and angiographic parameters at 6 months. All subjects will undergo assessments at 30 days and at 6 months. Additionally, all subjects will undergo a follow-up angiogram at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for catheter based treatment
* Single coronary lesion requiring treatment
* Lesion is accessible with stent device
* Completes informed consent for participation
* Stable condition (no symptoms of heart attack within 72 hours prior to treatment)

Exclusion Criteria:

* Normal lab values
* Previous treatment in the affected artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events(MACE). MACE defined as Cardiac Death, MI(Q-wave and Non Q-wave) and Rarget Vessel Revascularization (TVR) | 30 Days

SECONDARY OUTCOMES:
Clinical Outcome: MACE | 6 months
Clinical Outcome: Ischemia driven TVR | 6 months
Clinical Outcome: Ischemia driven Target LesionRevascularization(TLR) | 6 months
Clinical Outcome: Target Vessel Failure(TVF) | 6 months
Angiographic Outcome: Device Success defined as achievment of a final residual in-stent stenosis > 30%(by QCA) using the assigned device only | procedural
Angiographic Outcome: Lesion Success defined as attainment of a >30% residual in-stent stenosis (by QCA) using any percutaneous method | procedural
Angiographic Outcome: Procedural Success without the occurrence of cardiac death, Q-wave or Non Q-wave MI or repeat revascularization of the target lesion during the hospital stay. | hospital stay
Angiographic Outcome: Angiographic in-stent and in-segment binary restenosis rate(>/= 50% diameter stenosis) | at 6 months
Angiographic Outcome: In-stent, in-segment, proximal, and distal minimum lumen diameter(MLD)) | at 6 months
Angiographic Outcome: Angiographic in-stent late loss, defined as the difference between the post-procedural MLD and the follow-up MLD | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Instituto Dante Pazzanese de Cardioloigia, Sao Paulo, Brazil; Jeffery J Popma, MD, Principal Investigator — Brigham and Women's Hospital. Boston, Massachusetts, USA
Locations (3):
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto Do Coracao do Triangolo Mineiro, Uberlândia
- Johannes Gutenberg Universitat, Mainz, Germany

REFERENCES:
- [Result] Abizaid A, Popma JJ, Tanajura LF, Hattori K, Solberg B, Larracas C, Feres F, Costa Jde R Jr, Schwartz LB. Clinical and angiographic results of percutaneous coronary revascularization using a trilayer stainless steel-tantalum-stainless steel phosphorylcholine-coated stent: the TriMaxx trial. Catheter Cardiovasc Interv. 2007 Dec 1;70(7):914-9. doi: 10.1002/ccd.21279. PMID 18044791